CLINICAL TRIAL: NCT03069313
Title: A Single Arm Phase II Study of Oral Vitamin B12 for the Treatment of Aromatase Inhibitors (AI) Associated Musculoskeletal Symptoms in Women With Early Stage Breast Cancer
Brief Title: Vitamin B12 for Aromatase Inhibitors Musculoskeletal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Zeina Nahleh, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E15122
Record Dates: First submitted 2017-02-10; First posted 2017-03-03 (Actual); Results first posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Relief of Joint Pain
Keywords: Aromatase Inhibitor; Breast Cancer; Arthralgia; Musculoskeletal symptoms; Joint pain
MeSH Terms: conditions — Breast Neoplasms; Arthralgia | interventions — Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Vitamin B12 is to be taken sublingually on a daily basis for 90 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Oral Vitamin B12
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — Vitamin B12 2500 micrograms sublingually per day over the course of 90 days (+/- 10 days)

SUMMARY:
Significant Aromatase Inhibitor-associated toxicity, affects as many as 50% of patients with breast cancer leading to early discontinuation of this life-saving cancer treatment. No effective pharmacologic therapy has yet been identified for management of these symptoms, as many patients do not experience relief of symptoms with analgesic therapy. Vitamin B12, whether as injection or oral forms, has been used as a naturopathic product to provide relief for joint pain caused by arthritis. This effect has not been studied in the setting of Aromatase Inhibitor-Associated Musculoskeletal Symptoms (AIMSS).

DETAILED DESCRIPTION:
Primary Objectives:

a. To assess whether daily oral Vitamin B12 decreases average joint pain in women with aromatase inhibitor-associated musculoskeletal symptoms (AIMSS), as measured at baseline, 6 weeks and at 12 weeks by the modified Brief Pain Inventory Short Form (BPI-SF).

Secondary Objectives:

1. To investigate whether daily vitamin B12 improves functional quality of life as measured by the Functional Assessment of Cancer Therapy-Endocrine Scale (FACT-ES);
2. To explore the impact of treatment on serum inflammatory cytokine levels (C Reactive Protein) with 12 weeks of treatment between baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent and Pain level > 4 in the BPI scale,
* Stage I-III

Exclusion Criteria:

* <18 yrs
* Stage IV
* BPI Score <4
* Zubrod score >2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer patients
Enrollment: 41 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, Principal Investigator — Texas Tech University HSC El Paso

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: we needed at least a total of 30 patients to achieve more than 85% power to detect the differences in BPI-SF pain scores relative to baseline using a two tailed paired t-test with 5% level of significance. After accounting for 15% dropouts, we estimated to include at least 35 patients in the study.
Pre-assignment Details: IRB approved recruitment of 50 participants
Period: Overall Study
Arm/Group | Arm I
Started | 41
Completed | 36
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Average Joint Pain in Women With Aromatase Inhibitor-associated Musculoskeletal Symptoms (AIMSS) Compared to Baseline as Measured by the Brief Pain Inventory Short Form (BPI-SF).
Description: The Brief Pain Inventory - Short Form (BPI- SF) average pain score used. This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine" We expect at least 20% improvement in BPI-SF pain scores. Participants were asked to rate worst pain an average pain within the last 24 hours.
Time Frame: Baseline and 90 days (+/- 10 days)
Population: A total of forty-one patients were enrolled, five patients withdrew, leaving thirty-six patients to complete the study.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Arm I
Number analyzed (Participants) | 36
Percentage change | -33.8 (34.1)
Statistical Analysis 1: Comparison: Arm I; Test type: Other — Paired t-test; p < 0.0001, t-test, 1 sided

2. Secondary Outcome: Percentage Change in Worst Pain at the End of Treatment .
Description: Analysis of the data collected at baseline and at the end of treatment in the BPI-SF questionnaire. The Brief Pain Inventory - Short Form (BPI- SF) worst pain score used. This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine". Participants were asked to rate worst pain an average pain within the last 24 hours.
Time Frame: Baseline and 90 days (+/- 10 days)
Population: Postmenopausal women with ER+ breast cancer, stages I-III on aromatase inhibitors and musculoskeletal pain (average pain level > or=4 using BPI-SF)
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Arm I
Number analyzed (Participants) | 36
Percentage change | -23.03 (43.1)
Statistical Analysis 1: Comparison: Arm I; Test type: Other; p = 0.0003, t-test, 2 sided

3. Secondary Outcome: Percentage Change in Functional Quality of Life as Measured by the Functional Assessment of Cancer Therapy-Endocrine Scale (FACT-ES)
Description: All of the items in this questionnaire have a 5 scale rating, from not at all (0) to very much (4). Outcomes were measured pre and post treatment. Version 4 of the FACT-ES contains 3 subscales with seven questions: Physical Well-Being (PWB) (score range 0-28), Functional Well-Being (FWB) (score range 0-28), and Social and Well-Being (SWB) (score range 0-28); Emotional Well-Being (EWB) (score range 0-24) with six questions, and the Endocrine Symptom Subscale (ESS) (score range 0-76) containing 19 questions. For all subscale a higher score represents better quality of life.
Time Frame: Baseline and 90 days (+/- 10 days)
Population: postemneopausal women with ER + , Stages I-III breast cancer
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Arm I
Number analyzed (Participants) | 36
Percentage change
  SWB | 10.02 (27.7)
  EWB | 10.8 (38.6)
  PWB | 46.3 (62.5)
  FWB | 18 (45)
  ESS | 15.6 (19.6)
Statistical Analysis 1: Comparison: Arm I; Test type: Other — This analysis is comparing SWB before and after treatment; p = 0.133, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I; This analysis is comparing EWB before and after treatment; Test type: Other; p = 0.056, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm I; This analysis is comparing PWB before and after treatment; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm I; This analysis is comparing FWB before and after treatment; Test type: Other; p = 0.09, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm I; This analysis is comparing ESS before and after treatment; Test type: Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Percentage Change of Serum Levels of Vitamin B12, C-reactive Protein (CRP), Homoscyteine (HCys) and Methylmalonic Acid (MMA).
Description: Inflammatory markers were measured pre and post treatment.
Time Frame: Baseline and at 90 days (+/- 10 days)
Population: postmenopasual women receiving AI
Measure: Median (Standard Deviation); unit: Percentage change
Arm/Group | Arm I
Number analyzed (Participants) | 36
Percentage change
  B12 | 209.8 (191.3)
  CRP | 64.2 (298.5)
  HCys | -24.6 (19.75)
  MMA | -7.1 (81.65)

ADVERSE EVENTS:
Time Frame: 90 Days (+/- 10 days)
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 14/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=36)
dry mouth and nausea (Gastrointestinal disorders) | 14 (19)
blurred vision (Eye disorders) | 1 (1) — grade 1

LIMITATIONS AND CAVEATS:
Five of 41 participants did not complete the study medications and were not analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03069313/Prot_SAP_000.pdf